CLINICAL TRIAL: NCT05628805
Title: Theta Burst Stimulation to Improve Inhibitory Motor Physiology in Tourette Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Tourette Association of America (Other)
Responsible Party: Principal Investigator, Travis Larsh, Assistant Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-0747
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Tourette Syndrome; Tourette Syndrome in Children; Tourette Syndrome in Adolescence; Tourette Syndrome, Modifier of
MeSH Terms: conditions — Tourette Syndrome; Modifier, X-Linked, for Neurofunctional Defects

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- iTBS (Experimental): Each participant will have two separate study days in the TMS lab. On one day, the participant will receive active pre-SMA iTBS. On the other day, the patricipant will receive sham pre-SMA iTBS. The order that active versus sham is given will be randomized and the participant will be blinded. After each iTBS session, blinding assessment will be performed. To avoid contamination of results, a minimum of 5 days between study days will be required.
  Interventions: Device: iTBS
- Sham iTBS (Sham Comparator): Each participant will have two separate study days in the TMS lab. On one day, the participant will receive active pre-SMA iTBS. On the other day, the patricipant will receive sham pre-SMA iTBS. The order that active versus sham is given will be randomized and the participant will be blinded. After each iTBS session, blinding assessment will be performed. To avoid contamination of results, a minimum of 5 days between study days will be required.
  Interventions: Device: iTBS

INTERVENTIONS:
Device: iTBS — intermittent theta burst stimulation with TMS

SUMMARY:
Decades of Tourette Syndrome (TS) neuroimaging research has revealed abnormal cortical and subcortical motor system network, hypothesized to result from maladaptive plasticity. Repetitive transcranial magnetic stimulation ([r]TMS) is a promising technology that utilizes the concept of neuroplasticity to modulate brain circuits. TMS modulation has the distinct advantage in terms of its non-invasive nature. Furthermore, unique stimulation paradigms such as intermittent theta-burst repetitive TMS (iTBS) allows for short stimulation time (<3 min).

Using a sham-controlled protocol, the investigators propose modulating pre-SMA output using iTBS, based on our prior data of abnormal pre-SMA-mediated motor system regulation. hypothesize pre-SMA modulation results in increased pre-SMA-mediated motor inhibition. Enhancing these inhibitory measures with pre-SMA-iTBS provides the basis for improving inhibitory function in TS patients, leading to our long-term goal of neuro-stimulation to achieve clinical tic reduction.

ELIGIBILITY:
Inclusion Criteria:

Participants of any sex, race, or ethnicity meeting all criteria listed below will be included in the study:

1. Aged 10-21 years
2. Fluent in English
3. DSM-5 diagnosis of TS, confirmed by the clinical team
4. Able to participate in the informed consent process, provide voluntary informed consent/assent and provide a spontaneous narrative description of the key elements of the study.
5. Clinical stability: determined by a physician, no switch of psychotropic medications or increase in dosage in the last 14 days from TMS treatment start; no change in other therapeutic interventions in last 14 days from TMS treatment start.

Exclusion Criteria:

1. Any neurodevelopmental, psychiatric condition other than TS, ADHD, or OCD, or mild anxiety based on review of K-SADS. Note - if an exclusionary psychiatric diagnosis is suspected based on K-SADS, the research physician will follow up with the parent and referral will be made to psychology or psychiatry as appropriate.
2. Presence of metallic foreign bodies or implanted medical devices.
3. Not meeting inclusion criteria as described above
4. Non-fluency in English, as English is the language in the validated clinical questionnaires, and the participant must be able to understand real-time instructions from the study staff

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-02-16 (Estimated); Study Completion 2026-02-16 (Estimated)

PRIMARY OUTCOMES:
change in cortical silent period (cSP) | On the same day, we will assess change in cSP prior to active (or sham) iTBS treatment and immediately after iTBS treatment
  cSP is a biomarker of inhibitory motor physiology

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No